CLINICAL TRIAL: NCT03944395
Title: Assessing the Effectiveness and Feasibility of Voluntary Assisted Partner Notification Services in High HIV Burden Districts of Malawi: a Pragmatic, Non-Randomized Stepped-Wedge Study
Brief Title: Assessing the Effectiveness and Feasibility of Voluntary Assisted Partner Notification Services
Acronym: VAPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lighthouse Trust (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency); Elizabeth Glaser Pediatric AIDS Foundation (Other); Ministry of Health, Malawi (Other Government)
Responsible Party: Principal Investigator, Hannock Tweya, PhD, MSc, Director of Monitoring, Evaluation and Research, Lighthouse Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VAPN
Record Dates: First submitted 2018-07-16; First posted 2019-05-09 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: HIV Infections
Keywords: Active HIV Case finding; Partner Notification Services
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: A non-randomized, pragmatic, stepped-wedge study to be implemented in 80 Sites. The stepped wedge portion of the study will last 10 months (May - March 2018). Once all 80 sites are implementing standard of care (SOC) plus VAPN, the study will be extended an additional 3 months to assess any trends in declining yield from SOC plus VAPN index case testing services.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assisted Partner notification services (Other): Voluntary assisted partner notification (VAPN) services will be offered at facilities according to a stepped wedge design. Once VAPN services are activated at a facility, HIV positive individuals will be offered four options (3 voluntary assisted partner notification options and 1 standard of care option) for inviting their contacts, which they can choose to accept or decline.
  Interventions: Other: Assisted Partner Notification Services

INTERVENTIONS:
Other: Assisted Partner Notification Services — Three options for partner Notification services; contract referral, provider referral and dual referral

SUMMARY:
To evaluate effectiveness of voluntary assisted partner notification (VAPN) in real-world programmatic settings, a non-randomized, stepped wedge study in high volume facilities in 6 high HIV burden focus districts (Blantyre, Zomba, Chikwawa, Machinga, Mangochi and Lilongwe urban) is proposed. The primary objective is to compare the percentage of contacts tested during the standard of care (SOC) phase (i.e., using passive family referral services (FRS) index testing methodology) with the percentage of contacts tested during the SOC plus VAPN phase, by 1, 2, and 3 months after the initial contact with the index client. Assessment of feasibility will be achieved through documentation of operational lessons learned during implementation. Findings will contribute to ongoing policy discussions whether Malawi should adopt VAPN in its national HIV testing guidelines

DETAILED DESCRIPTION:
The over-arching goal of this study is to evaluate the effectiveness and feasibility of the voluntary assisted partner notification (VAPN) intervention in real-world programmatic settings in high burden facilities in 6 priority districts in Malawi.

The primary objective is to compare effectiveness of standard of care (SOC) (i.e., use of the family referral services (FRS)) with SOC plus VAPN in reaching contacts of index clients with HIV testing services. The percentage of contacts who receive HIV testing services within 1, 2, and 3 months of the initial offer of services to the index client will be compared between the SOC phase and the intervention phase (SOC plus VAPN).

Secondary objectives include:

1. To evaluate feasibility of implementing VAPN in real-world programmatic settings in high burden facilities in 6 priority districts in Malawi. Two key quantitative measures of feasibility will be used as follows:

   * What is the cumulative percentage of eligible index clients offered VAPN services by study end?
   * To what extent were the interventions implemented with fidelity? For example, a key measure of the fidelity of the Client Referral VAPN option is to assess what percentage of contacts, who did not return for their scheduled first appointment at the clinic, were subsequently traced according to the specified algorithm (i.e., up to 5 phone calls, and up to 2 home visits)?
2. To monitor trends in HIV diagnostic yield from SOC plus VAPN over time.

The study will include three options in additional to the FRS as part of the World Health organisation-recommended index testing approach. The first option is contract referral, in which the index client can choose to enter into a "contract" with the healthcare provider whereby he or she agrees to disclose their HIV status to all partners and refer them to HIV testing services (HTS) within a certain time frame. If the partners do not access HTS within this period, the providers will contact the partners directly to notify them that they may have been exposed to HIV; the providers will then offer voluntary HTS while maintaining the confidentiality of the index client. The second option is that of provider referral, in which the index client can choose to have the healthcare provider contact the client's partners directly, provide them with an appropriate health message, and offer them voluntary HTS, while maintaining the confidentiality of the index client. The third option is dual referral, in which the index client can choose that a trained provider sits with the client and his/her partner at a suitable time and location (usually a private room at the health facility) to provide support as they potentially test together or the index client discloses his/her HIV status with the provider offering voluntary HTS to the partner.

ELIGIBILITY:
Inclusion criteria:

Index clients:

* All index clients who are 18 years old or older (i.e., new positives, known positives not on treatment, and known positives who are on treatment), will be eligible for the study and eligible to receive VAPN services if informed consent is given.
* Index clients who are inpatients and pregnant women are eligible for inclusion in the study and in VAPN services if informed consent is given.

Contacts:

• All contacts of any age are eligible to be included in the study and eligible to receive HIV testing services according to Ministry of Health (MOH) guidelines. The age of consent to receive any component of HIV testing services in Malawi is 13. Prior to testing a contact (e.g., a child of an index case) who is <13 years old, for HIV, the guardian's consent is needed, per MOH guidelines.

Exclusion criteria:

Index clients

* Did not consent
* Aged <18 years old a
* Prisoners, Mentally disabled
* Intimate partner violence
* Cannot explain the three VAPN options (contract, referral, and dual referral) in a way that would result in true informed assent on the part of the client.

Contacts:

• There are no exclusion criteria for contacts to be included in the study or receive HIV testing services if they or their guardian desire services. Contacts who are <13 years old will not be contacted by phone under any VAPN contact outreach scenario.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1785 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-04-29 (Estimated); Study Completion 2020-04-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible index clients offered VAPN services | 10 months
  Number of eligible index clients who are offered VAPN divide by the number of all eligible index clients identified for enrolment

SECONDARY OUTCOMES:
Proportion of contacts who returned for HIV testing | 10 months
  Number of contacts who return for HIV testing divided by the number of contacts who are expected to return for HIV testing

OTHER OUTCOMES:
HIV Yield over time | 10 months
  Proportion of Contacts who tested HIV positive during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health Facilities, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Undecided